CLINICAL TRIAL: NCT02346929
Title: Comparison of Ultrasound-guided Hematoma Block and "Blind" Hematoma Block for Analgesia in Distal Radius Fractures
Brief Title: Hematoma Block for Distal Radius Fracture
Acronym: Hematoma Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Beatrice Hoffmann, ED Faculty, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000173
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Distal Radius Fracture
Keywords: Hematoma block; distal radius fracture reduction; ultrasound; ultrasound guided hematoma block; traditional hematoma block for analgesia; bupivacaine; pain reduction; wrist fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultrasound-guided hematoma block (Experimental): Patients in this arm will receive a bed-side ultrasound guided hematoma block with analgesia (0.25% bupivacaine)
  Interventions: Other: ultrasound guide
- traditional hematoma block (No Intervention): Patients in this arm will have the hematoma block of the distal radius fracture with no ultrasound for guidance with analgesia (0.25% bupivacaine)

INTERVENTIONS:
Other: ultrasound guide — Patients randomized to this arm will have the hematoma block of the distal radial fracture with the guidance of a bedside ultrasound
  Arms: ultrasound-guided hematoma block

SUMMARY:
The purpose of this study is to determine the efficacy of ultrasound guided hematoma block versus traditional "blind" hematoma block for analgesia in distal radius fracture reduction.

DETAILED DESCRIPTION:
Hematoma blocks are safe and effective in providing analgesia for fracture reduction1-4. They involve injecting lidocaine directly into the fracture line for analgesia. The physician aspirates blood prior to injection to confirm placement in the hematoma created by the fracture. However, the procedure can be technically difficult if the fracture line is difficult to palpate, for example, due to significant swelling or body habitus. Ultrasound has been shown to improve efficacy in other analgesic procedures such as peripheral nerve blocks5 and also in identifying fracture lines6. There have been case reports and case series which have shown the feasibility and effectiveness of ultrasound guided hematoma blocks for analgesia in patients undergoing reduction for distal radius fractures7,8. To our knowledge there are no randomized controlled trials comparing the use of ultrasound guided hematoma blocks versus traditional hematoma blocks in achieving analgesia for distal radius fracture reduction.

In this study, we will determine if ultrasound improves the efficacy of analgesia when performing hematoma blocks for reduction of distal radius fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years old presenting to the emergency department with complaint of distal radius fracture

Exclusion Criteria:

* High acuity/distress per the Attending ED physician
* Altered mental status or intoxication
* Aphasia, mental retardation, dementia, or insurmountable communication barrier
* Acute psychiatric illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction as indicated by Visual Analog Scale | 4 hours after initiation of study procedure
  Subjects will be surveyed on a Visual Analog Scale (VAS) on their pain during 4 points: prior to receiving hematoma block, after receiving hematoma block, during reduction and prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Hoffmann, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Furia JP, Alioto RJ, Marquardt JD. The efficacy and safety of the hematoma block for fracture reduction in closed, isolated fractures. Orthopedics. 1997 May;20(5):423-6. doi: 10.3928/0147-7447-19970501-11. PMID 9172249
- [Background] Alioto RJ, Furia JP, Marquardt JD. Hematoma block for ankle fractures: a safe and efficacious technique for manipulations. J Orthop Trauma. 1995 Apr;9(2):113-6. doi: 10.1097/00005131-199504000-00004. PMID 7776029
- [Background] Singh GK, Manglik RK, Lakhtakia PK, Singh A. Analgesia for the reduction of Colles fracture. A comparison of hematoma block and intravenous sedation. Online J Curr Clin Trials. 1992 Oct 1;Doc No 23:[3614 words; 43 paragraphs]. PMID 1343612
- [Background] Johnson PQ, Noffsinger MA. Hematoma block of distal forearm fractures. Is it safe? Orthop Rev. 1991 Nov;20(11):977-9. PMID 1749663
- [Background] Walker KJ, McGrattan K, Aas-Eng K, Smith AF. Ultrasound guidance for peripheral nerve blockade. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD006459. doi: 10.1002/14651858.CD006459.pub2. PMID 19821368
- [Background] Atkinson P, Lennon R. Use of emergency department ultrasound in the diagnosis and early management of femoral fractures. Emerg Med J. 2003 Jul;20(4):395. doi: 10.1136/emj.20.4.395. No abstract available. PMID 12835377
- [Background] Crystal CS, Miller MA, Young SE. Ultrasound guided hematoma block: a novel use of ultrasound in the traumatized patient. J Trauma. 2007 Feb;62(2):532-3. doi: 10.1097/01.ta.0000244398.89188.9c. No abstract available. PMID 17297348
- [Background] Kiely PD, O'Farrell D, Riordan J, Harmon D. The use of ultrasound-guided hematoma blocks in wrist fractures. J Clin Anesth. 2009 Nov;21(7):540-2. doi: 10.1016/j.jclinane.2009.01.008. No abstract available. PMID 20006267